CLINICAL TRIAL: NCT01603381
Title: The Effect of Family History on Insomnia During Sobriety in Alcoholics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhajit Chakravorty, Staff Physician, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01257
Record Dates: First submitted 2012-02-03; First posted 2012-05-22 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I (Experimental): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Monitor Only (M.O.) (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Behavioral management of insomnia
  Arms: CBT-I

SUMMARY:
The investigators intend to assess the following:

* the efficacy of CBTi in treating insomnia during recovery,
* does a family history of alcoholism moderate the insomnia symptoms,
* does an improvement in insomnia lead to a decrease in impulsivity.

DETAILED DESCRIPTION:
The primary goals of this pilot study are the following:

a) to assess for the difference in improvement insomnia, after 8 weeks of treatment with recommended CBTi, in Veterans with alcohol dependence during early recovery,

The secondary goals include the following:

1. to assess for any change in the alcohol consumption indices between the groups after 8 weeks of CBTi,
2. to assess for change in psychiatric symptoms of mood and anxiety across the groups,
3. to assess for differences in insomnia in subjects, with and without a first degree family history of alcohol dependence,
4. to evaluate for any change in impulsivity-related measure with insomnia treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of insomnia currently
2. DSM IV diagnosis of alcohol dependence within the past year
3. Not in acute alcohol withdrawal and within a year of sobriety from alcoholism
4. Patients with moderate-severe sleep apnea compliant on their PAP device
5. Can speak, understand and print in English.
6. Is capable of giving written informed consent.

Exclusion Criteria:

1. Dependence on psychoactive substance (excluding alcohol, nicotine and cannabis) in the past 12 months, or evidence of chronic opiate use.
2. Unstable/serious psychiatric condition e.g. schizophrenia, bipolar disorder.
3. Unstable or serious medical/neurologic illness
4. Severe cognitive impairment
5. Untreated moderate - severe obstructive sleep apnea

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index total score | 8 weeks.
  There will be post-treatment follow up at 3 months and 6 months.

SECONDARY OUTCOMES:
Time Line Follow Back measure | 8 weeks.
  There will be post-study follow-up at 3 months and 6 months also.

CONTACTS AND LOCATIONS:
Overall Officials: Subhajit Chakravorty, M.D., Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Chakravorty S, Morales KH, Arnedt JT, Perlis ML, Oslin DW, Findley JC, Kranzler HR. Cognitive Behavioral Therapy for Insomnia in Alcohol-Dependent Veterans: A Randomized, Controlled Pilot Study. Alcohol Clin Exp Res. 2019 Jun;43(6):1244-1253. doi: 10.1111/acer.14030. Epub 2019 Apr 29. PMID 30912860